CLINICAL TRIAL: NCT04680429
Title: A Phase I, Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study and Food Effect Study of Oral RP7214, a DHODH Inhibitor, in Healthy Volunteers
Brief Title: A Single and Multiple Ascending and Food Effect Study of RP7214, a DHODH Inhibitor in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rhizen Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RP7214-2002
Record Dates: First submitted 2020-12-17; First posted 2020-12-23 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Healthy Volunteers
Keywords: DHODH
MeSH Terms: interventions — RP7214

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RP7214, Single and multiple doses (Experimental): In Part 1 up to 3 cohorts with single ascending doses of RP7214 at 100 mg QD, 200 mg QD and 400 mg QD.
  In Part 2 up to 2 cohorts with multiple ascending doses of RP7214 at 200 mg BID, 400 mg BID.
  Interventions: Drug: RP7214
- Placebo, Single and multiple doses (Placebo Comparator): In Part 1 up to 3 cohorts and in Part 2 up to 2 cohorts with matching placebo to RP7214 tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RP7214 — Participants will receive single and multiple ascending doses of RP7214
  Arms: RP7214, Single and multiple doses
Drug: Placebo — Participants will receive single and multiple ascending doses of matching placebo
  Arms: Placebo, Single and multiple doses

SUMMARY:
This is a randomized, double-blind study to evaluate the safety, tolerability and PK of single and multiple ascending oral doses of RP7214. The relative bioavailability in fed and fasting conditions will also be evaluated for RP7214. The study comprises three parts; Part 1: Single ascending dose, Part 2: Multiple ascending dose and Part 3: Food effect.

DETAILED DESCRIPTION:
There are three escalating cohorts in SAD part and two escalating cohorts in MAD part. In each cohort, six eligible healthy volunteers will be randomized to receive either RP7214 or placebo in 2:1 ratio. Within each cohort, two sentinel subjects (RP7214 and Placebo) will be dosed first for assessment of safety and tolerability. The safety data of at least 48 hrs will be reviewed to confirm safety of sentinel subjects after which the remaining four subjects will be dosed. Food effect study is a randomized, 2-treatment, 2-period, 2-sequence, crossover study in 12 HVs.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects willing and able to provide informed consent for the trial
2. Male and non-childbearing female subjects aged 18 to 55 years
3. Healthy subjects as determined by pre-study medical history, vitals, physical examination and 12-lead ECG, and clinical laboratory tests within the normal reference ranges or clinically acceptable to investigator
4. Non-tobacco user/non-smokers or ex-smokers defined as someone who has stopped smoking cigarettes for at least 6 months.
5. Negative screen for drugs of abuse and alcohol at screening and on admission.
6. Body mass index (BMI) between 18.0 and 32.0 kg/m2 inclusive.
7. A male subject who is able to procreate should agree to use one of the accepted contraceptives and agree to refrain from donating sperm for at least 3 months after dosing; and should not father a child during this period.
8. Female subjects should be of non-childbearing potential.
9. Willing and able to understand the nature of this study, comply with the study procedures as required by the study protocol.

Exclusion Criteria:

1. Subjects with evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies) at the time of screening.
2. Positive screen for hepatitis-B surface antigen (HBsAg), antibodies to the hepatitis C (HCV) or antibodies to the human immunodeficiency virus (HIV) 1 and 2.
3. Subjects who received or are on Covid-19 directed prophylaxis (e.g. chloroquine or hydroxychloroquine) in last two weeks or 5x half-lives of the drug, whichever is shorter, prior to dosing.
4. Subjects participating in another clinical study or use of any investigational product in last 30 days or 5x half-lives of the drug, whichever is shorter, prior to dosing.
5. Pregnant or lactating females.
6. Clinically significant abnormalities in physical examination and/or in laboratory tests (including hematology and chemistry panels, urinalysis) as assessed by the Investigator.
7. Donation or loss of 400 mL or more of blood within eight (8) weeks prior to initial dosing, or longer if required by local regulations/procedures.
8. Concomitant disease or condition that could interfere with the conduct of the study, or for which the treatment could interfere with the conduct of the study, or that would in the opinion of investigator, pose an unacceptable risk to the subject in this study.
9. Inability or unwillingness to comply with study and/or follow-up procedures outlined in the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2021-07-17 (Actual); Study Completion 2021-07-19 (Actual)

PRIMARY OUTCOMES:
Assessments of Adverse Events (AEs) | Day1 - day15

SECONDARY OUTCOMES:
RP7214 Cmax | 0, 0.25, 0.5, 1, 2, 4, 6, 8 and 12 hrs post dose
  Maximum Observed Plasma Concentration
RP7214 Tmax | 0, 0.25, 0.5, 1, 2, 4, 6, 8 and 12 hrs post dose
  Time for maximum plasma concentration
RP7214 t½ | 0, 0.25, 0.5, 1, 2, 4, 6, 8 and 12 hrs post dose
  Terminal half-life
RP7214 AUC0-inf | 0, 0.25, 0.5, 1, 2, 4, 6, 8 and 12 hrs post dose
  Area under the plasma concentration time curve from zero extrapolated to infinite time

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rhizen Investigational Site, Las Vegas, Nevada
  - Rhizen Investigational Site, Fargo, North Dakota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nair A, Barde PJ, Routhu KV, Viswanadha S, Veeraraghavan S, Pak S, Peterson JA, Vakkalanka S. A first in man study to evaluate the safety, pharmacokinetics and pharmacodynamics of RP7214, a dihydroorotate dehydrogenase inhibitor in healthy subjects. Br J Clin Pharmacol. 2023 Mar;89(3):1127-1138. doi: 10.1111/bcp.15562. Epub 2022 Nov 1. PMID 36217901